CLINICAL TRIAL: NCT05864027
Title: Oral Health Recovery: A Peer-Delivered Oral Health Intervention for Individuals With Psychiatric Disabilities
Brief Title: Oral Health Recovery Group
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Blue Cross Blue Shield of Michigan Foundation (Other)
Responsible Party: Principal Investigator, Adrienne Lapidos, Clinical Assistant Professor, Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00219880
Record Dates: First submitted 2023-04-12; First posted 2023-05-18 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Oral Health; Dental Care; Psychiatric Diagnosis
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer-led Oral Health Recovery educational group (Experimental)
  Interventions: Behavioral: Peer-led Oral Health Recovery Group
- Educational Video (Active Comparator)
  Interventions: Behavioral: Educational Video about Oral Health

INTERVENTIONS:
Behavioral: Peer-led Oral Health Recovery Group — The interactive Oral Health Recovery group will be centered around the tailored materials previously developed, with topics such as "it's never too late to make a change," "oral health and whole health," "taking care of your teeth," and "going to the dentist."
  Arms: Peer-led Oral Health Recovery educational group
Behavioral: Educational Video about Oral Health — The video comparison will be pulled from Toothflix 2.0 Patient Education DVD Series, which are patient education videos developed by the American Dental Association.
  Arms: Educational Video

SUMMARY:
The aim of the study is to test a brief, peer-led group-based oral health educational intervention - called the "Oral Health Recovery Group" - designed for individuals with psychiatric disabilities.

DETAILED DESCRIPTION:
Participants at each site will obtain either: a) a Peer-led Oral Health Recovery educational group, representing the primary intervention; or b) viewing of an educational video about oral health, representing the comparison intervention. After participating in either condition, an onsite Peer staff member will offer to help the participant make a dentist appointment. They will follow up with the participant as needed for a two-month period to help arrange dental care and follow up on any dental self-care goals established by the participant, such as purchasing toothpaste with fluoride.

ELIGIBILITY:
Inclusion Criteria:

* An adult member/consumer with the selected site (JIMHO or Washtenaw CMH)
* Ability to understand and willingness to read a consent terms handout and discussion
* Participant must understand/read/speak English

Exclusion Criteria:

* Not a member/consumer with the site
* Not able to understand and/or not willing to read consent terms handout
* Does not understand/read/speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Average subject-level change between pre- and post-surveys | 2 months
  To analyze process data generated by the peers, a custom web-based Peer Encounter Form will be employed using Qualtrics Survey Software. Peers will complete encounter forms after each group and follow up. Fields include time spent, unique and total encounters, topics covered, participant engagement, and any knowledge of participants' seeking out or utilizing dental care.
  The primary analyses will compare the change in total scores on an oral health knowledge questionnaire and an oral health confidence/activation questionnaire based primarily on the transtheoretical model of change. These comparisons will be conducted as a comparison of the average subject-level improvements between pre- and post-surveys ("change scores") between the primary intervention (peer-led Oral Health Recovery Group) and the comparator video intervention.

SECONDARY OUTCOMES:
Odds ratio of participants who reported seeking dental care | 2 months
  Odds ratio comparing the odds of seeking care in the two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne Lapidos, PhD, Principal Investigator — University of Michigan Medical School, Psychiatry
Locations (2):
- United States (2):
  - Justice in Mental Health Organization (JIMHO), Lansing, Michigan
  - Community Mental Health (Towner), Ypsilanti, Michigan

IPD SHARING:
Plan to Share IPD: No